CLINICAL TRIAL: NCT03645993
Title: Early Onset Alzheimer's Disease Genomic Study
Acronym: TGen
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 017-176
Record Dates: First submitted 2018-07-27; First posted 2018-08-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Early-Onset Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Plasma Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early-Onset Alzheimer's disease: Patients ages 45-60 with Early-Onset Alzheimer's disease
  Interventions: Genetic: Genetic Testing
- Negative Control: Family members of patients with Early-Onset Alzheimer's disease who have consented to the study.

INTERVENTIONS:
Genetic: Genetic Testing — A one time blood sample will be taken.
  Groups: Early-Onset Alzheimer's disease

SUMMARY:
The purpose of this study is to collect samples from patients with Early-Onset Alzheimer's disease (AD) and their immediate family members for molecular analysis. Samples will be studied in order to understand how molecular changes in the body are related to the development of the disease. Researchers will study your DNA and RNA in order to help doctors diagnose, treat, and monitor people at risk of developing Early-Onset AD in the future.

DETAILED DESCRIPTION:
About 50 people will be asked to take part in this study at this location. This will include participants with early-onset AD and their parents and siblings. Participants will be asked to: Sign this consent form or have a Legally Authorized Representative sign and provide the participant' health history. The study staff will review the participant's medical history and test results to see if the participant can be part of this study, The study staff will need to know any over-the-counter or prescription drugs, vitamins, or herbs taken by the participant. The study staff will discuss what is required to be part of this study. Participants cannot take part in this study if they have: Family history of early or late-onset Alzheimer's disease, Uncontrolled concurrent illness including psychiatric illness or situations that would limit compliance with the study requirements or the ability to willingly give written or verbal consent. If the participant agrees to take part in this study, one 8mL blood sample (about 2 teaspoons) will be collected from them. If the participant is receiving a clinically indicated blood draw, the blood collections for this study will occur at the same time. Participants may be required to have a research-specific blood draw if they are not scheduled for a blood draw during a regularly scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early-onset Alzheimer's disease based on the NIA-AA diagnostic criteria as determined by the clinician. (Those patients with severe dementia due to Alzheimer's disease or who have impaired decisional capacity, may participate only if their legally authorized representative gives their consent.)
* Male and female patients ≥40 and ≤65 years of age.
* Parents and siblings of the participant with Alzheimer's disease.

Exclusion Criteria:

* Family history of early or late-onset Alzheimer's disease.
* Uncontrolled concurrent illness including psychiatric illness or situations that would limit compliance with the study requirements or the ability to willingly give written or verbal informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of early-onset Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Biomarkers found in blood | 2 years
  Blood will be taken so that tests can be run to locate a biomarker that will help to diagnose and treat early-onset Alzheimer's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White AT&T Memory Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No